CLINICAL TRIAL: NCT02520453
Title: Randomised, Double-blind, Phase II Trial of Adjuvant Durvalumab or Placebo for Completely Resected Esophageal Squamous Cell Carcinoma Previously Treated With Neoadjuvant Concurrent Chemoradiotherapy
Brief Title: Adjuvant Durvalumab for Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Mu Sun, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-06-166
Record Dates: First submitted 2015-08-04; First posted 2015-08-11 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Durvalumab (Experimental): Durvalumab 20 mg/Kg IV Q 4 weeks for 1 year, or until disease relapse or unacceptable toxicity
  Interventions: Drug: Durvalumab
- Placebo (Placebo Comparator): Placebo Q 4 weeks for 1 year, or until disease relapse or unacceptable toxicity
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Durvalumab
  Arms: Durvalumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
Adjuvant Durvalumab vs Placebo for 1 year after complete resection of esophageal cancer following neoadjuvant CCRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous esophageal cancer, irrespective of PD-L1 status
* The enrolment should be done during the time interval from 20 days to 56 days after complete resection after neoadjvuant CCRT (no residual tumor after operation)
* Clinical tumor stage before neoadjuvant CCRT should be T3-4N0M0 or T1-4N1-3M0
* Available tumor specimen for biomarker analysis acquired before neoadjuvant CCRT or at operation

Exclusion Criteria:

* Other PD-1 or PD-L1 inhibitors history
* Mean QT interval corrected for heart rate (QTc) ≥470 ms using Bazett's correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Mu Sun, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, MA, South Korea